CLINICAL TRIAL: NCT04447911
Title: Effects of the SGLT2 Inhibitor Empagliflozin in Patients With Euvolemic and Hypervolemic Hyponatremia - a Multicentric Randomized Double-blind Placebo-controlled Trial (the EMPOWER Study)
Brief Title: Effects of the SGLT2 Inhibitor Empagliflozin in Patients With Euvolemic and Hypervolemic Hyponatremia
Acronym: EMPOWER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Luzerner Kantonsspital (Other); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMPOWER study
Record Dates: First submitted 2020-06-10; First posted 2020-06-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Hyponatremia; SIADH; Liver Failure; Kidney Failure
MeSH Terms: conditions — Hyponatremia; Inappropriate ADH Syndrome; Liver Failure; Renal Insufficiency | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Multicentric prospective randomized double-blind placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental): Empagliflozin (Jardiance)® 25mg per os once daily for 30 days
  Interventions: Drug: Empagliflozin 25 MG
- Placebo (Placebo Comparator): Placebo (Lactose tablet) per os once daily for 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Empagliflozin 25mg per os once daily for 30 days
  Arms: Empagliflozin
Drug: Placebo — Placebo per os once daily for 30 days
  Arms: Placebo

SUMMARY:
Hyponatremia is the most common electrolyte derangement occurring in hospitalized patients. It is usually classified as hypovolemic, euvolemic or hypervolemic. The most common aetiology of euvolemic hyponatremia is the syndrome of inappropriate antidiuresis (SIAD). Hypervolemic hyponatremia is common in patients with congestive heart failure (CHF) (10-27%) and liver cirrhosis (up to approximately 50%). In SIAD, the regulation of arginine vasopressin (AVP) secretion is impaired which leads to free water retention. In CHF and liver cirrhosis, the effective arterial blood volume is decreased leading to non-osmotic baroreceptor mediated AVP release and consecutive free water retention.

Current treatments of euvolemic and hypervolemic hyponatremia, including the most used treatment fluid restriction, are of limited efficacy. Sodium-Glucose-Co-Transporter 2 (SGLT2) inhibitors reduce glucose reabsorption in the proximal tubule, resulting in glucosuria and consecutive osmotic diuresis. A placebo-controlled randomized trial of our group has shown that a short-term, i.e. a 4-days administration of the SGLT2 inhibitor empagliflozin (Jardiance)® in addition to fluid restriction was effective in increasing the serum sodium concentration in 87 patients with SIAD-induced hyponatremia. The effect of empagliflozin (Jardiance)® without additional fluid restriction is however not yet known. Large randomized controlled trials have shown that SGLT2 inhibitors reduced hospitalization for heart failure in patients with, and more recently without type 2 diabetes. No studies have investigated the effect of SGLT2 inhibitors in hypervolemic hyponatremia.

To evaluate the effect of empagliflozin (Jardiance)® in eu- and hypervolemic hyponatremia, a randomized placebo-controlled study is needed.

ELIGIBILITY:
Inclusion Criteria:

- chronic eu- OR hypervolemic non hyperosmolar (<300 mOsm/kg) hyponatremia (heparin plasma sodium <135 mmol/L on day of inclusion)

Exclusion Criteria:

* known hypersensitivity or allergy to class of drugs or the investigational product,
* severe symptomatic hyponatremia in need of treatment with 3% NaCl-solution or in need of intensive/intermediate care treatment at time of inclusion
* clinical hypovolemia
* Severe reduction of eGFR <20 mL/min/1,73 m2 (KDIGO G4 and G5) or end stage renal disease
* Chronic liver insufficiency with Child Pugh Score ≥10 or decompensated liver cirrhosis (jaundice, hepatorenal syndrome, encephalopathy, bleeding, …)
* Hepatic impairment defined as aspartate transaminase (AST) or alanine transaminase (ALT) >3x the upper limit of normal (ULN); or total bilirubin >2x ULN at time of enrolment
* uncontrolled hypothyroidism
* uncontrolled adrenal insufficiency
* systolic blood pressure <90mmHg
* contraindication for lowering blood pressure
* diabetes mellitus type 1 or pancreatic diabetes mellitus
* treatment with SGLT2 inhibitors, lithium chloride, vaptans, demeclocycline or urea on inclusion day
* severe immunosuppression (leucocytes <2 G/l)
* peripheral arterial disease stage III-IV of the Fontaine Classification
* fasting or other reasons preventing medication intake
* previous enrolment into the current study
* participation in another intervention study
* pregnancy, breastfeeding, intention to become pregnant during the course of the study or lack of safe contraception.
* end of life care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in average daily area under curve (AUC) for serum sodium concentration | 4 days
  Change in average daily AUC for serum sodium concentration
Long-term serum sodium change (before/after treatment) | 30 days
  Absolute change in serum sodium concentration from baseline to end of treatment

SECONDARY OUTCOMES:
Impact intervention on bodyweight | 30 days
  change of bodyweight
Impact intervention on blood pressure | 30 days
  change of blood pressure
Course of serum sodium level | 30 days
  Course of serum sodium level
Change of plasma osmolality | 30 days
  Change of plasma osmolality
Change of urinary osmolality | 30 days
  Change of urinary osmolality
Change of plasma urea | 30 days
  Change of plasma urea
Change of urinary urea | 30 days
  Change of urinary urea
Change of plasma uric acid | 30 days
  Change of plasma uric acid
Change of urinary uric acid | 30 days
  Change of urinary uric acid
Change of plasma creatinin | 30 days
  Change of plasma creatinin
Change of urinary creatinin | 30 days
  Change of urinary creatinin
Change of plasma potassium | 30 days
  Change of plasma potassium
Change of urinary potassium | 30 days
  Change of urinary potassium
Change in plasma copeptin | 30 days
  Change in plasma copeptin
Change in plasma aldosterone | 30 days
  Change in plasma aldosterone
Change in plasma renin | 30 days
  Change in plasma renin
Change in plasma MR-proANP | 30 days
  Change in plasma MR-proANP
Change in plasma NT-proBNP | 30 days
  Change in plasma NT-proBNP
Change in plasma CTX | 30 days
  Change in plasma CTX
Change in plasma P1NP | 30 days
  Change in plasma P1NP
Occurence of thirst | 30 days
  Occurence of thirst
Occurence of headache | 30 days
  Occurence of headache
Occurence of vertigo | 30 days
  Occurence of vertigo
Occurence of nausea | 30 days
  Occurence of nausea
Change in general well-being | 30 days
  Change in general well-being according to visual analogue scale
Change in quality of life | 30 days
  change in quality of life according to EQ-5D-5L questionnaire
Change in cognitive impairment | 30 days
  Change in cognitive impairment measured with the MoCa test
Change in visual attention | 30 days
  Change in visual attention measured with the trail making test
Change in neuromuscular impairment | 30 days
  Change in neuromuscular impairment measured with the timed up and go test
Change in grip strength | 30 days
  Change in grip strength measured with a hand dynamometer
Occurence of falls | 30 days
  Occurence of falls
Occurence of fractures | 30 days
  Occurence of fractures
Length of hospital stay | 30 days
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Julie Refardt, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (6):
- University Hospital of Würzburg, med. Poliklinik, Würzburg, Germany
- Erasmus Universität Medisch Centrum Rotterdam, Department of Internal Medicine, Rotterdam, Netherlands
- Switzerland (4):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - University Hospital Basel, Basel
  - Spitalzentrum Biel, Biel
  - Kantonsspital Luzern, Lucerne

IPD SHARING:
Plan to Share IPD: Yes